CLINICAL TRIAL: NCT02640937
Title: Biofilm Formation Increases Treatment Failure in Staphylococcus Epidermidis Device-related Osteomyelitis in Human Patients
Brief Title: Biofilm Formation in Staphylococcus Epidermidis Associated Implant Infections
Status: Completed | Type: Observational
Sponsor: BG Unfallklinik Murnau (Other)
Responsible Party: Principal Investigator, Dr. Mario Morgenstern, Specialist in Orthopedic Surgery, BG Unfallklinik Murnau
Other Study IDs: 12063
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Staphylococcal Infections
Keywords: Staphylococcus epidermidis; biofilm formation; antibiotic resistance; Orthopaedic device related infections; risk factor
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial samples from orthopaedic device realted infections
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orthopaedic device related infections: Inclusion Criteria:
  * infections after fracture fixation or prosthetic joint surgery
  * Affected bone or joint: Long bones of the lower extremity; hip joint, knee joint;
  * Bacterial growth of S. epidermidis at the site of interest
  * Written consent
  * Age: 18 and older

SUMMARY:
This was a prospective study performed between November 2011 and September 2013. Patients with a confirmed S. epidermidis infection after fracture fixation or prosthetic joint infection were included. Exclusion criteria included infections involving external fixation pins, infections without any implanted hardware and culture positive patients not displaying any clinical sign of infection. The following surgical parameters were documented: affected bone or joint; type of implant; time between implantation of the device and onset of symptoms. Personal characteristics and patients'health status were also documented. Any revision surgeries involving the site of interest and all isolated pathogens were recorded throughout the course of treatment and follow-up.

A follow up examination was performed an average of 26 months after discharge. Primary outcome at follow up was cure. Cure was define by the authors as: missing local (at site of interest) or systemic signs of infection, terminated surgical and systemic therapy and restoration of joint or limb function.

At the first surgical procedure after enrolment, at least four deep bone biopsies were taken from the interface between implant and affected bone. Identification and antibiotic susceptibility testing of all growth was performed. Multi-drug-resistance (MDR) was defined according to the definitions of the European Committee of Antimicrobial Susceptibility Testing (EUCAST). Biofilm formation was analysed and quantified in microtitre plate assays according to protocol of Stepanovic et al.(see references).

DETAILED DESCRIPTION:
This was a prospective study performed between November 2011 and September 2013. All patients provided informed written consent prior to inclusion in the study. Inclusion criteria were deep S. epidermidis infections after fracture fixation or prosthetic joint surgery. Fracture fixation infections includes fractures involving the long bones as well as the pelvis and the spine. Bacterial growth at the site of interest in combination with either pseudarthrosis, implant-loosening/failure or local and systemic signs of surgical site infection were required for inclusion. Exclusion criteria included infections involving external fixation pins, infections without any implanted hardware and culture positive patients not displaying any clinical sign of infection.

Upon entry into the study, the following surgical parameters were documented: affected bone or joint; type of implant; time between implantation of the device and onset of symptoms. Personal characteristics were also documented and included: gender; age; body mass index (BMI); smoker/non-smoker; overall medical condition (Charlson comorbidity index); and chronic immunosuppressive conditions (Diabetes mellitus, chronic alcoholism, Child's class C cirrhosis, neoplasia, transplantation, AIDS and steroid medication). Any revision surgeries involving the site of interest and all isolated pathogens were recorded throughout the course of treatment and follow-up.

A follow up examination was performed an average of 26 months after discharge. Primary outcome at follow up was cure. Cure was define by the authors as: missing local (at site of interest) or systemic signs of infection and terminated surgical and systemic therapy.

At the first surgical procedure after enrolment, at least four deep bone biopsies were taken from the interface between implant and affected bone. The tissue samples were placed in a sterile container with thioglycollate liquid medium (bioMérieux, Hazelwood, MO, USA). The samples were cultured for ten days at 37°C and examined each day macroscopically. Any growth was inoculated onto a blood agar plate (bioMérieux, Hazelwood, MO, USA) for further growth and subsequent identification. In all cases, additional swabs and soft tissue samples may have been taken as per clinical routine, however, only samples adjacent to the implant were used for diagnosis in this study.

Identification and antibiotic susceptibility testing of all growth was performed using a Vitek2 (bioMerieux Vitek Inc, Hazelwood, MO, USA). Multi-drug-resistance (MDR) was defined according to the definitions of the European Committee of Antimicrobial Susceptibility Testing (EUCAST). Oxacillin resistance was used as an indicator for methicillin resistant S. epidermidis (MRSE).

Biofilm formation was analysed and quantified in microtitre plate assays according to the well-established protocol of Stepanovic et al.(see references). This method traditionally assigns isolates to one of four categories: non-biofilm-formers and weak, moderate or strong biofilm-formers.

The key variables with regards to bacterial phenotype were: biofilm formation; methicillin resistance; and multidrug resistance. The primary outcome measure was whether the infection was "cured" or not. Primary outcome parameters were calculated as a function of all patients for whom data was complete. Statistical comparison was restricted to the lower extremity cohort since the other patients are not scored for many of the functional outcome measures and as such incomplete.

Univariate logistic regression models were used to determine the influence of each prognostic factor (obesity, smoking, diabetes mellitus, chronic immune suppression, open fracture (initially), early onset infection, biofilm formation, methicillin resistance, MDR and Charlson comorbidity index) on cure. P-values <0.05 were considered signiﬁcant. Statistical analyses were performed using SAS software (Version 9.2; Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* infections after fracture fixation or prosthetic joint surgery
* Affected bone or joint: Long bones of the lower extremity; hip joint, knee joint;
* Bacterial growth of S. epidermidis at the site of interest
* Written consent
* Age: 18 and older

Exclusion Criteria:

* no prove of bacterial growth at site of interest
* missing consent
* infections involving external fixation pins, infections without any implanted hardware.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic device related infection involving longbones of the lower extermity
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2011-11; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cure | 24 month
  Cure was define by the authors as: missing local (at site of interest) or systemic signs of infection and terminated surgical and systemic antibiotic therapy. All Parameters had to be positive to fulfill the outcome parameter "cure".If one of the mentioned parameters was negative, outcome was defined as "not cured". Local signs of infection were defined as the appearance of: redness, tenderness, swelling or persisting wound drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Morgenstern, M.D., Principal Investigator — BGUnfallklinik Murnau
Locations (1):
- BG Unfallklinik Murnau, Murnau am Staffelsee, Bavaria, Germany

REFERENCES:
- [Background] Stepanovic S, Vukovic D, Hola V, Di Bonaventura G, Djukic S, Cirkovic I, Ruzicka F. Quantification of biofilm in microtiter plates: overview of testing conditions and practical recommendations for assessment of biofilm production by staphylococci. APMIS. 2007 Aug;115(8):891-9. doi: 10.1111/j.1600-0463.2007.apm_630.x. PMID 17696944
- [Derived] Post V, Harris LG, Morgenstern M, Mageiros L, Hitchings MD, Meric G, Pascoe B, Sheppard SK, Richards RG, Moriarty TF. Comparative Genomics Study of Staphylococcus epidermidis Isolates from Orthopedic-Device-Related Infections Correlated with Patient Outcome. J Clin Microbiol. 2017 Oct;55(10):3089-3103. doi: 10.1128/JCM.00881-17. Epub 2017 Aug 9. PMID 28794175